CLINICAL TRIAL: NCT04781257
Title: Early Risk Assessment in TB contactS by New Diagnostic tEsts
Brief Title: Early Risk Assessment in Household Contacts (≥10 Years) of TB Patients by New Diagnostic Tests in 3 African Countries
Acronym: ERASE-TB
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Michael Hoelscher (Other)
Collaborators: European and Developing Countries Clinical Trials Partnership (EDCTP) (Other Government)
Responsible Party: Sponsor-Investigator, Michael Hoelscher, Professor Dr., Ludwig-Maximilians - University of Munich
Organization: Ludwig-Maximilians - University of Munich (Other)
Other Study IDs: LMU-IMPH-AIDA-03
Record Dates: First submitted 2020-12-21; First posted 2021-03-04 (Actual); Last update posted 2023-11-28 (Actual); Status verified 2023-11

CONDITIONS: Tuberculosis
Keywords: Tuberculosis; Latent Tuberculosis; Pulmonary Tuberculosis; Case-Control Studies; Disease Transmission, Infectious; Blood Specimen Collection; Urine Specimen Collection; Sputum; Diagnostic Techniques and Procedures; Biomarkers; Interferon-gamma Release Tests; Mass Chest X-ray; Radiography; Respiratory Function Tests; Spirometry; Artificial Intelligence; Transcriptome; Biological Specimen Banks; Models, Theoretical; Housing; Family Characteristics; Africa South of the Sahara; Zimbabwe; Mozambique; Tanzania
MeSH Terms: conditions — Tuberculosis; Latent Tuberculosis; Tuberculosis, Pulmonary; Communicable Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Urine, Serum, Plasma, Full blood, Peripheral blood mononuclear cells (PBMCs), Sputum
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Household contacts with co-prevalent/incipient TB: Household contacts diagnosed with active TB at baseline/during the study period
  Interventions: Diagnostic Test: New test candidates
- Household contacts staying healthy: Household contacts without active TB who remain healthy throughout the study
  Interventions: Diagnostic Test: New test candidates

INTERVENTIONS:
Diagnostic Test: New test candidates — The following new diagnostic tests will be done after the completion of the study with the samples (blood, sputum, urine) and data (digital X-ray) obtained during the study period:
  CAD4TB / qXR Xpert Ultra® FLOW-TB TAM-TB 4RISK and COR Cepheid 3-gene signature cartridge BioMérieux ISIT TB blood transcription signature assay Multiplex LSHTM in-house host biomarker assay TB Screen biosignature SeroSelect
  Retrospective testing of participants' samples and data acquired during the study period, differentiated between participants with co-prevalent/incipient TB and participants staying health throughout the trial

SUMMARY:
The ERASE - TB study will be conducted in order to fill a critical unmet need for tuberculosis control. Persons who are in contact with an infectious TB case may become infected themselves. Among those who are infected, most will stay healthy but some will develop TB themselves.

These people would benefit from preventive treatment, which would also stop TB from being spread to other persons.

The problem currently is that it is impossible to determine with certainty who would require preventive treatment, and who will remain healthy. Out of 100 persons exposed to an infectious TB patient, only 2 will go on to have TB according to a study in Vietnam, but there are no good tests available to identify those with a risk for TB disease. Treating 100 persons to prevent 2 cases of TB is not effective, so preventive treatment is not used in adults and adolescents in Tanzania, Mozambique and Zimbabwe, where this study will be conducted, but also in many other settings.

The ERASE - TB project will evaluate a number of newly developed diagnostic tests, to see which of those will be able to predict TB in persons at risk, and therefore steer preventive treatment well.

For this, the investigators will invite 2,100 household contacts (HHC) of infectious TB patients, who are at least 10 years old, into the study. Everyone will be examined initially, and again in regular intervals, for 1.5 to 2 years; and whenever the participants will present with symptoms that could indicate that they develop TB.

At every visit, the investigators will perform an X-ray and take some blood and urine samples to perform new candidate tests. At the first/baseline visit, all household contacts without TB will undergo a spirometry to evaluate their pulmonary function.

If someone is unwell, the investigators will also examine sputum for the presence of TB bacilli. In the end, the investigators will then be able to say who of the persons in the study developed TB, and who remained healthy. From all samples taken at different timepoints, the investigators will then determine which test found TB early, and clearly distinguished between persons developing TB, and persons who would remain healthy .

ELIGIBILITY:
Inclusion Criteria:

TB index case:

* Aged at least 18 years
* Having at least one other person living in the household aged ≥10 years
* Written informed consent to conduct socio-economic and clinical questionnaire, to provide a sputum sample for culture and sequencing, and to approach the household members.
* Recently diagnosed with active pulmonary TB within the last 4 weeks
* Has taken less than 7 daily doses of anti-TB treatment since diagnosis; ensuring a positive culture can still be obtained
* Able to spontaneously produce sputum
* Sputum microscopy positive in Ziehl-Neelsen or Auramine-O staining of ideally 2+ or higher, but at least 1+ on the IUATLD/WHO scale, OR (in case no sputum microscopy done) GeneXpert positive, at least TB "medium"
* A firm home address, maintained unchanged for the last 6 months, that is accessible to visiting

Household Contact:

* Aged at least 10 years
* Written informed consent for study participation, including HIV testing, and home visits by the study team for follow-up (for minors <18 yr.: consent of the parent/guardian, assent of the participant)
* Recent (in the last 4 weeks), substantial exposure to an infectious TB case in the household, defined as sleeping at least 3/7 nights in the same household
* If HIV negative: not on preventive therapy (preventive therapy is not an exclusion criterion for HIV positive persons)

Exclusion Criteria:

Household Contact

* Circumstances that raise doubt on free, uncoerced informed consent (e.g. in a mentally handicapped person)
* Prisoners
* Recent treatment for active TB, completed within the last 30 days OR on current TB treatment for active TB.

Min Age: 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: TB index cases will be recruited at the primary health care clinics where the patient is receiving TB treatment. Household contacts have substantial recent exposure to the TB index case in the household (defined as sleeping at least 3/7 nights in the same household in the last 4 weeks).
Sampling Method: Non-Probability Sample
Enrollment: 2100 (Estimated)
Dates: Start 2021-03-01 (Actual); Primary Completion 2024-04-30 (Estimated); Study Completion 2024-04-30 (Estimated)

PRIMARY OUTCOMES:
Sensitivity and specificity of new diagnostics to diagnose co-prevalent TB against a clinica/microbiological reference standard case definition | Co-prevalent TB disease can be diagnosed at Baseline (Month 0)
  to determine sensitivity and specificity of new diagnostics for diagnosing TB earlier with a special focus on subclinical disease.
  New diagnostics will be evaluated against a reference standard for classification of presence of, or development of TB disease in a person exposed to a source case; with the following possibilities:
  * Co--prevalent symptomatic TB
  * Co--prevalent subclinical TB
  * Minimal TB, with incident TB during follow-up
  * Remained healthy
Evaluation of novel diagnostics for detection of developing, minimal TB against a clinica/microbiological reference standard case definition | TB disease can be diagnosed through study completion, up to Month 24
  to evaluate novel diagnostics for detection of developing, minimal TB that would cause infectious disease in the future.
  For reference standard case classification, see 1.
Enhancement of diagnostic performance by simulating testing algorithms coupled with a risk estimate from a mathematical model | TB disease can be diagnosed through study completion, up to Month 24
  to enhance diagnostic performance by simulating testing algorithms coupled with a risk estimate from a mathematical model For reference standard case classification, see 1.

SECONDARY OUTCOMES:
M.tb infection status as measured by an immunological assay | through study completion, up to Month 24
  M.tb infection status as measured by an immunological assay:
  * M.tb infected at baseline
  * M.tb uninfected at baseline through to end of study
  * Change of M.tb infection status from negative (baseline) to positive during follow-up
Classification of cases of co-prevalent or incident TB; through M.tb isolate sequencing and comparison with the source case isolate | through study completion, up to Month 24
  Classification of cases of co-prevalent or incident TB; through M.tb isolate sequencing and comparison with the source case isolate:
  * Secondary, infected by source case - defined timepoint of infection
  * Other, unknown source of infection - unknown timepoint of infection
Assessment of the proportion of HHC (without co-prevalent TB) with abnormal pulmonary function at baseline | Spirometry will be done only at baseline
  to assess the proportion of HHC (without co-prevalent TB) with abnormal pulmonary function at baseline, the type and severity of impairments, the relationship between pre-existing abnormal pulmonary function and incident TB (and the changes in pulmonary function measured by spirometry after incident TB and TB treatment completion).

OTHER OUTCOMES:
To explore elements shaping adoption of new TB detection technologies among asymptomatic members of community (sub-study I) | August 2021 to February 2022
  In-depth qualitative interviews will be conducted to understand how new technologies could support screening and follow-up of household contacts.

CONTACTS AND LOCATIONS:
Overall Officials: Theodora Mbunda, MD, PhD, Principal Investigator — National Institute of Medical Research - Mbeya Medical Research Centre; Denise F Banze, MD, Principal Investigator — Instituto Nacional de Saúde (INS); Junior Mutsvangwa, MD, Principal Investigator — Biomedical Research & Training Institute (BRTI)
Locations (3):
- Instituto Nacional de Saúde (INS) Centro de Investigação e Treino em Saúde da Polana Caniço, Maputo, Mozambique
- NIMR - Mbeya Medical Research Centre, Mbeya, Tanzania
- Biomedical Research & Training Institute (BRTI), Harare, Zimbabwe

IPD SHARING:
Plan to Share IPD: Undecided
Accordance with EU General Data Protection Regulation and local data protection law needs to be worked out.

REFERENCES:
- [Background] Drain PK, Bajema KL, Dowdy D, Dheda K, Naidoo K, Schumacher SG, Ma S, Meermeier E, Lewinsohn DM, Sherman DR. Incipient and Subclinical Tuberculosis: a Clinical Review of Early Stages and Progression of Infection. Clin Microbiol Rev. 2018 Jul 18;31(4):e00021-18. doi: 10.1128/CMR.00021-18. Print 2018 Oct. PMID 30021818
- [Background] Fox GJ, Nhung NV, Sy DN, Hoa NLP, Anh LTN, Anh NT, Hoa NB, Dung NH, Buu TN, Loi NT, Nhung LT, Hung NV, Lieu PT, Cuong NK, Cuong PD, Bestrashniy J, Britton WJ, Marks GB. Household-Contact Investigation for Detection of Tuberculosis in Vietnam. N Engl J Med. 2018 Jan 18;378(3):221-229. doi: 10.1056/NEJMoa1700209. PMID 29342390
- [Background] Swindells S, Ramchandani R, Gupta A, Benson CA, Leon-Cruz J, Mwelase N, Jean Juste MA, Lama JR, Valencia J, Omoz-Oarhe A, Supparatpinyo K, Masheto G, Mohapi L, da Silva Escada RO, Mawlana S, Banda P, Severe P, Hakim J, Kanyama C, Langat D, Moran L, Andersen J, Fletcher CV, Nuermberger E, Chaisson RE; BRIEF TB/A5279 Study Team. One Month of Rifapentine plus Isoniazid to Prevent HIV-Related Tuberculosis. N Engl J Med. 2019 Mar 14;380(11):1001-1011. doi: 10.1056/NEJMoa1806808. PMID 30865794
- [Derived] Marambire ET, Banze D, Mfinanga A, Mutsvangwa J, Mbunda TD, Ntinginya NE, Celso K, Kallenius G, Calderwood CJ, Geldmacher C, Held K, Appalarowthu T, Riess F, Panzner U, Heinrich N, Kranzer K; ERASE-TB Consortium. Early risk assessment in paediatric and adult household contacts of confirmed tuberculosis cases by novel diagnostic tests (ERASE-TB): protocol for a prospective, non-interventional, longitudinal, multicountry cohort study. BMJ Open. 2022 Jul 19;12(7):e060985. doi: 10.1136/bmjopen-2022-060985. PMID 36427173
- See also: WHO Global Tuberculosis Report 2019 — https://www.who.int/publications/i/item/9789241565714
- See also: Consensus Meeting Report: Development of a Target Product Profile (TPP) and a framework for evaluation for a test for predicting progression from tuberculosis infection to active disease — https://apps.who.int/iris/handle/10665/259176